CLINICAL TRIAL: NCT00642837
Title: Health - Related Quality of Life in Patients With Rheumatic Diseases Taking Tramadol 37.5mg/Acetaminophen 325mg Tablets ; Multicenter, Open-label, Prospective, Observational Study
Brief Title: A Study on Health - Related Quality of Life in Patients With Rheumatic Diseases Taking Tramadol 37.5mg/Acetaminophen 325mg Tablets
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014803
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatic Diseases
Keywords: Health-Related Quality of Life; KEQ-5D; Sleep disturbance; Sleep quality; SF-1; Pain intensity; Pain relief; Tramadol; Acetaminophen
MeSH Terms: conditions — Rheumatic Diseases; Parasomnias; Sleep Initiation and Maintenance Disorders; Pain | interventions — Ultracet

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (9):
- 001
  Interventions: Drug: Tramadol/acetaminophen
- 002
  Interventions: Drug: Tramadol/acetaminophen
- 003
  Interventions: Drug: Tramadol/acetaminophen
- 004
  Interventions: Drug: Tramadol/acetaminophen
- 005
  Interventions: Drug: Tramadol/acetaminophen
- 006
  Interventions: Drug: Tramadol/acetaminophen
- 007
  Interventions: Drug: Tramadol/acetaminophen
- 008
  Interventions: Drug: Tramadol/acetaminophen
- 009
  Interventions: Drug: Tramadol/acetaminophen

INTERVENTIONS:
Drug: Tramadol/acetaminophen — Osteoarthritis, flexible dose depending on patients' pain relief
  Groups: 002
Drug: Tramadol/acetaminophen — Post surgical neurophatic pain, flexible dose depending on patients' pain relief
  Groups: 008
Drug: Tramadol/acetaminophen — Post traumatic neuropathic pain, flexible dose depending on patient pain relief
  Groups: 009
Drug: Tramadol/acetaminophen — Spinal Cord Injury, flexible dose depending on patients' pain relief
  Groups: 005
Drug: Tramadol/acetaminophen — Failed Back Surgery Syndrome,flexible dose depending on patients' pain relief
  Groups: 006
Drug: Tramadol/acetaminophen — Diabetic Neuropathy, flexible dose depending on patients' pain relief
  Groups: 003
Drug: Tramadol/acetaminophen — Post stroke pain, flexible dose depending on patients' pain relief
  Groups: 007
Drug: Tramadol/acetaminophen — Low back pain, flexible dose depending on patients' pain relief
  Groups: 001
Drug: Tramadol/acetaminophen — Post Herpetic Neuralgia, flexible dose depending on patients' pain relief
  Groups: 004
Drug: Tramadol/acetaminophen — Complex Regional Pain Syndrome, flexible dose depending on patients' pain relief
  Groups: 006

SUMMARY:
The objective of this observational study is to assess improvement of quality of life in the patients who are administered Tramadol 37.5mg/Acetaminophen 325mg tablets for 10~14 weeks according to the investigator's discretion in clinical practice.

DETAILED DESCRIPTION:
Recently the concerns about the Health-Related Quality of Life (HRQOL) have been increasing especially in chronic diseases. Rheumatic disease is a chronic disease, which can result in a functional disability and impaired HRQOL. Because of this chronic pain, patients with rheumatic disease have lower scores on HRQOL than general population. A several studies have indicated Ultracet as an add-on treatment to nonsteroidal antiinflammatory drugs(NSAIDs) for osteoarthritis(OA) pain, fibromyalgia pain and chronic low back pain significantly improved HRQOL, compared with placebo. We will use the KEQ-5D (a Korean version of the EQ-5D which is a health related quality of life questionnaire) to assess HRQOL. The KEQ-5D has been shown to be effectively sensitive in several rheumatic conditions. The study hypothesis is that the quality of life will be improved after Tramadol 37.5mg/Acetaminophen 325mg tablets administration in outpatients who need Tramadol 37.5mg/Acetaminophen 325mg tablets administration at the investigator's discretion. This is a multicenter, open-label, prospective, observational study to compare HRQOL using Korean version of EQ-5D before and after the treatment with Tramadol 37.5mg/Acetaminophen 325mg tablets and to assess the correlation among each measurement. Observational Study - No investigational drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatism who have moderate-to-severe pain
* Patients who have not been administered Ultracet or tramadol over the last one month
* Patients who have signed a consent form indicating that they understand the purpose of and procedures required for the study (For minors between 12 and 20 years old, the patients' legally acceptable representatives' signature is also required.)

Exclusion Criteria:

* Patients who have experienced failure of tramadol therapy or discontinued Tramadol because of adverse events
* Patients with impaired physical function or disease which may cause drug absorption anomaly, excess storage and metabolic or elimination disorder
* Patients who meet any of the prohibitions of tramadol or acetaminophen
* Hypersensitive to active ingredients of the study drug
* Addicted to drugs acting on central nervous system including alcohol, hypnotics, centrally acting analgesics, opiates and psychotropics, serious respiratory depression (the study drug may cause mild respiratory depression)
* Patients with head injury and brain lesion who have the risk of decreased meantal awareness
* Patients who are taking an MAO inhibitor or discontinued it no more than 2 weeks ago
* Patients with peptic ulcer and severe hematological anomaly
* Patients with severe hepatic impairment, renal impairment or cardiac dysfunction
* Patients with aspirin-induced asthma (asthmatic attacks induced by nonsteroidal anti-inflammatory drug)
* Patients with epilepsy which is not controlled by a drug
* Patients who are pregnant or of childbearing potential during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rheumatism who have moderate-to-severe pain
Sampling Method: Probability Sample
Enrollment: 982 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
KEQ-5D: Korean Version of EQ-5D which assess the health related quality of life of patient | baseline and week 12

SECONDARY OUTCOMES:
Pain relief | baseline & week 12
Pain intensity | baseline & week 12

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.